CLINICAL TRIAL: NCT04942522
Title: Application of Probiotic PS128 (Lactobacillus Plantarum, PS128) in Children With Autism Spectrum Disorder (ASD)
Brief Title: Application of Probiotic PS128 in Children With ASD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Yan Hao (Other)
Responsible Party: Sponsor-Investigator, Yan Hao, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S313
Record Dates: First submitted 2021-06-02; First posted 2021-06-28 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Autism Spectrum Disorder
Keywords: ASD; probiotics
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASD children A (Experimental): Participants received probiotics PS128 [6×10^10 CFU(colony forming unit)/capsule} one capsule orally twice daily for 8 weeks. After a washout period (4 weeks), they then received placebo(450mg/capsule) one capsule orally twice daily for 8 weeks. Stool, urine and blood specimen will be collected at baseline, week 8, week 12 and week 20.
  Interventions: Biological: probiotics PS128; Drug: placebo (Microcrystalline cellulose )
- ASD children B (Experimental): Participants received placebo(450mg/capsule) one capsule orally twice daily for 8 weeks. After a washout period (4 weeks), they then received probiotics PS128(6×10^10 CFU/capsule) one capsule orally twice daily for 8 weeks. Stool, urine and blood specimen will be collected at baseline, week 8, week 12 and week 20.
  Interventions: Biological: probiotics PS128; Drug: placebo (Microcrystalline cellulose )

INTERVENTIONS:
Biological: probiotics PS128 — 6×10^10 CFU/capsule
Drug: placebo (Microcrystalline cellulose ) — 450 mg/capsule

SUMMARY:
The purpose of this study is to explore the role of probiotics PS128 in improving gastrointestinal dysfunction and core behavioral symptoms in children with ASD, and investigate the underlying etiological mechanisms of ASD.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo screening period to determine eligibility for study entry. Participants who meet the eligibility requirements will be randomized in a double-blind manner(participant and investigator) in a 1:1 ratio to probiotics PS128 group or placebo group. Each patient acts as his or her own control, and they receive both the study drug as well as the placebo. After a washout period, the participants will be switched throughout to different treatments（probiotics placebo group or PS128 group）.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2-5 years with ASD from Tongji hospital (both boys and girls);
2. meets Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and ADOS-2 diagnostic criteria;
3. No significant abnormalities on head MRI or EEG;
4. If psychotropic medication is required during the project, the psychiatrist must confirm that medication is stable during this period (no change in dose or type of medication);
5. Willing to provide samples such as blood, urine and feces.

Exclusion Criteria:

1. Take antibiotics or antifungal drugs within 15 days prior to the project.
2. Take probiotic products within 30 days prior to the project.
3. Have acute diarrhea within 30 days prior to the project.
4. Start taking new psychotropic medication within 15 days prior to the project.
5. Have severe hearing, visual or motor impairment.
6. Accompany with other mental behavioral disorders, such as schizophrenia, bipolar disorder.
7. A history of Rett syndrome, chromosomal, inherited metabolic disorders and other significant somatic disorders.
8. A history of organic gastrointestinal disorders (e.g., gastroesophageal reflux, food allergies, inflammatory bowel disease), history of intestinal surgery, intestinal obstruction, intestinal perforation, intestinal bleeding, multi-organ failure, and severe immunodeficiency disorders
9. Have a special diet (e.g., gluten-free diet, casein-free diet, ketogenic diet, etc.)
10. Co-morbidities in children with ASD were documented and discussed in detail by two or more behavioral developmental behaviorists, and children with ASD who required immediate rehabilitation or neurological analogs for co-morbidities were not allowed to enter this study.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2023-06-06 (Estimated); Study Completion 2023-10-06 (Estimated)

PRIMARY OUTCOMES:
change in Autism Diagnostic Observation Scale (ADOS) | Baseline, 8 weeks, 12 weeks and 20 weeks
  The ADOS consists of a series of structured and semi-structured tasks that involve social interaction between the examiner and the person under assessment. The examiner observes and identifies segments of the subject's behavior and assigns these to predetermined observational categories. Categorized observations are subsequently combined to produce quantitative scores for analysis and diagnostic classification of ASD. Children at or above predetermined cutoff lines are considered to be positive for ASD. The assessment will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.
change in Social Responsiveness Scale (SRS) | Baseline, 8 weeks, 12 weeks and 20 weeks
  The SRS is a 65-item rating scale with standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total scores results are as follows:
  0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment The assessment will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.
Change in Social Communication Questionnaire (SCQ) | Baseline, 8 weeks, 12 weeks and 20 weeks
  The SCQ is a 40-item survey where each question is a 'yes' or 'no' answer. The total possible range of scores is 0-39 (verbal children) or 0-33 (non-verbal children) with higher scores indicative of greater frequency of symptoms. The assessment will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.
Change in the Autism Behavior Checklist (ABC) | Baseline, 8 weeks, 12 weeks and 20 weeks
  ABC is a scale used for nonadaptive behaviors created to screen and indicate the probability of a diagnosis of autism. The questionnaire including 57 items related to five areas: sensorial, relational, use of body and objects, and social skills. Scale score> 67 strongly suggests the presence of autism. The assessment will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.
Change in the Childhood Autism Rating Scale (CARS) | Baseline, 8 weeks, 12 weeks and 20 weeks
  CARS assesses the child on a scale from 1 to 4 in each of 15 dimensions or symptoms. A total score of at least 30 strongly suggests the presence of autism. Children with score between 30 and 36 have mild-to-moderate autism while those with score between 37 and 60 have severe autism. The assessment will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.
Change in Gesell developmental scale | Baseline, 8 weeks, 12 weeks and 20 weeks
  The Gesell developmental scale mainly measures five areas: adaptive behavior, gross motor, fine motor, Language behavior, personal-social behavior, the evaluation finally calculates the developmental quotient (DQ) of each area. Diagnostic criteria: DQ is more than or equal to 86 is normal, DQ is marginal between 76 and 85, DQ is mild mental retardation between 55 and 75, DQ is moderate mental retardation between 40 and 54, DQ is severe mental retardation between 25 and 39, and DQ is less than or equal to 25 is extremely severe mental retardation. The assessment will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.
Change in frequency of child behavioral problems | Baseline, 8 weeks, 12 weeks and 20 weeks
  Child behavioral problems will be assessed using the Externalizing scale of the Child Behavior Checklist (CBCL) for Ages 1.5-5. The Externalizing scale measures child attention problems and aggressive behaviors using 24 items rated by parents based on child performance during the previous two months with a 3-point -type scale. The study will use the CBCL 1.5-5 for all families whose children will be between three to six years old. Lower scores suggest fewer behavioral problems. The assessment will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.
Change in frequency of ASD symptoms | Baseline, 8 weeks, 12 weeks and 20 weeks
  ASD symptoms will be assessed using the Chinese version of the Autism Treatment Evaluation Checklist (ATEC), which comprise four subscales to measure child speech/language/communication, sociability, sensory/cognitive awareness, and health/physical/behavior. The scale has 77 items that are scored by parents. The health/physical/behavior subscale is rated using a 0 (not a problem)-to-3 (serious problem) point scale, whereas the other three subscales are rated using a 0 (not true)-to-2 (very true) point scale. Higher scores represent more ASD symptoms. The assessment will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.
change in gastrointestinal symptoms among children with ASD | Baseline, 8 weeks, 12 weeks and 20 weeks
  Assessment will be conducted for the Rome IV diagnoses of cyclic vomiting, functional vomiting, functional dyspepsia, and/or functional constipation. The presence or absence of meeting criteria for the Rome IV diagnoses will be coded as a binary variable (true/false) to represent resolution of symptoms. The assessment will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.

SECONDARY OUTCOMES:
Cytokine Analysis | Baseline, 8 weeks, 12 weeks and 20 weeks
  Interleukin, Tumor necrosis factor and chemokines will be measured in patient peripheral blood. The analysis will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.
Evaluate changes of type, number and structural composition of gut microorganisms in children with ASD. | Baseline, 8 weeks, 12 weeks and 20 weeks
  Stool routine and 16S-rRNA to evaluate gut microorganisms. The analysis will be conducted before and after each intervention, namely baseline, 8 weeks, 12 weeks and 20 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Hao, PhD, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Data involves children's privacy.

REFERENCES:
- [Background] Elsabbagh M, Divan G, Koh YJ, Kim YS, Kauchali S, Marcin C, Montiel-Nava C, Patel V, Paula CS, Wang C, Yasamy MT, Fombonne E. Global prevalence of autism and other pervasive developmental disorders. Autism Res. 2012 Jun;5(3):160-79. doi: 10.1002/aur.239. Epub 2012 Apr 11. PMID 22495912
- [Background] Fombonne E. Epidemiology of pervasive developmental disorders. Pediatr Res. 2009 Jun;65(6):591-8. doi: 10.1203/PDR.0b013e31819e7203. PMID 19218885
- [Background] Xu G, Strathearn L, Liu B, O'Brien M, Kopelman TG, Zhu J, Snetselaar LG, Bao W. Prevalence and Treatment Patterns of Autism Spectrum Disorder in the United States, 2016. JAMA Pediatr. 2019 Feb 1;173(2):153-159. doi: 10.1001/jamapediatrics.2018.4208. PMID 30508021
- [Background] Bailey A, Le Couteur A, Gottesman I, Bolton P, Simonoff E, Yuzda E, Rutter M. Autism as a strongly genetic disorder: evidence from a British twin study. Psychol Med. 1995 Jan;25(1):63-77. doi: 10.1017/s0033291700028099. PMID 7792363
- [Background] Ronald A, Hoekstra RA. Autism spectrum disorders and autistic traits: a decade of new twin studies. Am J Med Genet B Neuropsychiatr Genet. 2011 Apr;156B(3):255-74. doi: 10.1002/ajmg.b.31159. Epub 2011 Jan 13. PMID 21438136
- [Background] de la Torre-Ubieta L, Won H, Stein JL, Geschwind DH. Advancing the understanding of autism disease mechanisms through genetics. Nat Med. 2016 Apr;22(4):345-61. doi: 10.1038/nm.4071. PMID 27050589
- [Background] Grafodatskaya D, Chung B, Szatmari P, Weksberg R. Autism spectrum disorders and epigenetics. J Am Acad Child Adolesc Psychiatry. 2010 Aug;49(8):794-809. doi: 10.1016/j.jaac.2010.05.005. Epub 2010 Jul 3. PMID 20643313
- [Background] Lord C, Risi S, Lambrecht L, Cook EH Jr, Leventhal BL, DiLavore PC, Pickles A, Rutter M. The autism diagnostic observation schedule-generic: a standard measure of social and communication deficits associated with the spectrum of autism. J Autism Dev Disord. 2000 Jun;30(3):205-23. PMID 11055457
- [Background] Frazier TW, Klingemier EW, Beukemann M, Speer L, Markowitz L, Parikh S, Wexberg S, Giuliano K, Schulte E, Delahunty C, Ahuja V, Eng C, Manos MJ, Hardan AY, Youngstrom EA, Strauss MS. Development of an Objective Autism Risk Index Using Remote Eye Tracking. J Am Acad Child Adolesc Psychiatry. 2016 Apr;55(4):301-9. doi: 10.1016/j.jaac.2016.01.011. Epub 2016 Feb 4. PMID 27015721
- [Background] Lai MC, Lombardo MV, Auyeung B, Chakrabarti B, Baron-Cohen S. Sex/gender differences and autism: setting the scene for future research. J Am Acad Child Adolesc Psychiatry. 2015 Jan;54(1):11-24. doi: 10.1016/j.jaac.2014.10.003. Epub 2014 Oct 16. PMID 25524786
- [Background] Shattuck PT, Durkin M, Maenner M, Newschaffer C, Mandell DS, Wiggins L, Lee LC, Rice C, Giarelli E, Kirby R, Baio J, Pinto-Martin J, Cuniff C. Timing of identification among children with an autism spectrum disorder: findings from a population-based surveillance study. J Am Acad Child Adolesc Psychiatry. 2009 May;48(5):474-483. doi: 10.1097/CHI.0b013e31819b3848. PMID 19318992
- [Background] Reinhardt VP, Wetherby AM, Schatschneider C, Lord C. Examination of sex differences in a large sample of young children with autism spectrum disorder and typical development. J Autism Dev Disord. 2015 Mar;45(3):697-706. doi: 10.1007/s10803-014-2223-6. PMID 25189824
- [Background] Rose AJ, Rudolph KD. A review of sex differences in peer relationship processes: potential trade-offs for the emotional and behavioral development of girls and boys. Psychol Bull. 2006 Jan;132(1):98-131. doi: 10.1037/0033-2909.132.1.98. PMID 16435959